CLINICAL TRIAL: NCT04801342
Title: Neurocognitive Outcome of Conformal Whole Brain Radiotherapy With Bilateral or Unilateral Hippocampal Avoidance Plus Memantine for Brain Metastases: A Phase II Single Blind Randomized Trial
Brief Title: Neurocognitive Outcome of Bilateral or Unilateral Hippocampal Avoidance WBRT With Memantine for Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901084MINA
Record Dates: First submitted 2019-04-28; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Malignant Neoplasm to Brain
Keywords: Brain Metastases; Hippocampal Avoidance Whole Brain Radiotherapy; Neurocognitive function
MeSH Terms: conditions — Brain Neoplasms | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Unilateral Hippocampal Avoidance WBRT with Memantine (Experimental): Conformal whole brain radiotherapy with unilateral hippocampal avoidance and Concurrent use of Memantine HCL
  Interventions: Radiation: Conformal Whole Brain Radiotherapy with Unilateral Hippocampal Avoidance; Drug: Memantine Hydrochloride
- Bilateral Hippocampal Avoidance WBRT with Memantine (Active Comparator): Conformal whole brain radiotherapy with bilateral hippocampal avoidance and Concurrent use of Memantine HCL
  Interventions: Radiation: Conformal Whole Brain Radiotherapy with Bilateral Hippocampal Avoidance; Drug: Memantine Hydrochloride

INTERVENTIONS:
Radiation: Conformal Whole Brain Radiotherapy with Unilateral Hippocampal Avoidance — Conformal Whole Brain Radiotherapy 30 Gy in 10 fractions with Unilateral Hippocampal Avoidance using Intensity modulated radiotherapy, Volumetric arc therapy, or Tomotherapy
  Other Names: Unilateral HA-WBRT
  Arms: Unilateral Hippocampal Avoidance WBRT with Memantine
Radiation: Conformal Whole Brain Radiotherapy with Bilateral Hippocampal Avoidance — Conformal Whole Brain Radiotherapy 30 Gy in 10 fractions with Bilateral Hippocampal Avoidance using Intensity modulated radiotherapy, Volumetric arc therapy, or Tomotherapy
  Other Names: Bilateral HA-WBRT
  Arms: Bilateral Hippocampal Avoidance WBRT with Memantine
Drug: Memantine Hydrochloride — Start from day 1 of WBRT orally for 24 weeks and escalating doses over the first 4 weeks
  Other Names: Memantine

SUMMARY:
Brain metastases are the most common brain tumors in adults. It is estimated that around 10-30% of cancer patients would develop brain metastases during the course of their illness.

Whole brain radiotherapy (WBRT) is the treatment of choice for the majority of patients with brain metastases. WBRT yields high radiologic response rate (27~56%) and is effective in rapid palliation of neurologic symptoms as well as prolongs time to neurocognitive function decline caused by intracranial lesions. By using conventional fractionation, more than one- third of patients developed late neurocognitive toxicity while memory impairment was the most common symptom. The incidence is even higher when a formal and sensitive neurocognitive assessment was prospectively evaluated. With more long-term survivors nowadays, it has become increasingly important to minimize neurocognitive function decline and maintain quality of life in patients with brain metastasis.

The function of hippocampus is cooperation in learning, consolidation and retrieval of information and essential for formation of new memories. Bilateral and unilateral radiation injury of the hippocampus is known to alter learning and memory formation. Several preclinical studies support the hypothesis of hippocampus-mediated cognitive dysfunction by ionizing radiation. Clinical studies show increase in radiation dose to hippocampus is associated with subsequent neurocognitive function impairment in adult and pediatric patients. Furthermore, the result of phase III randomized trials suggested hippocampal avoidance plus Memantine significantly reduce the risk of neurocognitive impairment at 6 months from 68.2% in control arm with standard WBRT to 59.5% in experimental arm. In the investigator's prior investigation, patients received conformal WBRT with bilateral hippocampal avoidance also had significant less declines in verbal memory at 6 months.

Previous studies showed the right and left hippocampus exert different neurocognitive functions. Several retrospective studies also demonstrated that the radiation dose to the left hippocampus is more related to neurocognitive impairment. Planning study and investigation showed that by avoiding the left hippocampus alone, the radiation dose to the spared unilateral hippocampus is further decreased. In present study, a single blind randomized phase II trial is designed to investigate the effectiveness of neurocognitive function preservation using conformal WBRT with bilateral or unilateral hippocampal avoidance and memantine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of non-hematopoietic malignancy and radiographic evidence of brain metastases
* Patients with brain metastasis outside a 5-mm margin around either hippocampus on gadolinium contrast enhanced MRI obtained within 30 days prior to registration
* Patients with brain metastasis who have not been or will not be treated with SRS, or have received SRS for ≤ 5 intracranial metastatic lesion(s)
* No evidence of diffuse leptomeningeal metastasis on gadolinium- enhanced MRI within 30 days prior registration
* Age ≥ 20 years
* Karnofsky Performance Status ≥ 60%
* Life expectancy of ≥ 6 months.
* Women of childbearing potential and male participants must practice adequate contraception
* Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion Criteria:

* Prior radiotherapy to brain or radiosurgery to > 5 intracranial metastatic lesion(s) or the biological equivalent dose in 2-Gy fractions was greater than 7.3Gy to 40% of the volume of bilateral hippocampus from prior radiosurgery
* Serum creatinine > 2.0 mg/dL within 30 days prior registration
* Serum urea nitrogen > 20 mg/dL within 30 days prior registration
* Contraindication to MR imaging such as implanted metal devices or foreign bodies, severe claustrophobia
* Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

  1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
  2. Transmural myocardial infarction ≤ 6 months prior to registration
  3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
  4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
  5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  7. Uncontrolled psychiatric disorder
* Will receive any other investigational agent or chemotherapy during WBRT
* Current use of Memantine HCL or Allergy to Memantine HCL
* Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic
* Pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVLT-R) memory score | At 6 months after WBRT
  Decline in Hopkins Verbal Learning Test-Revised (HVLT-R) memory score (sum of total recall and recognition index) from baseline to 6 months after the start of conformal whole brain radiotherapy (WBRT) with bilateral or unilateral hippocampal avoidance for multiple brain metastases. HVLT-R Total recall raw scores ranged from 0 to 36, recognition index ranged from 0 to 12. The higher the score indicated better short term memory preservation

SECONDARY OUTCOMES:
Neurocognitive function by a standardized neurocognitive battery Hopkins Verbal Learning Test-Revised (HVLT-R) | at 1, 2, 4, 6, 9, 12 months after WBRT, and then every 3 months until date of death from any cause, assessed up to 24 months
  Evaluate neurocognitive function by a standardized neurocognitive battery Hopkins Verbal Learning Test-Revised (HVLT-R) with Total recall score (range from 0 to 36), delayed recall score (range from 0 to 12) and recognition index (range from 0 to 12). The higher the score indicated better short term memory preservation.
Neurocognitive function by a standardized neurocognitive battery Trail Making Test Part A & B | at 1, 2, 4, 6, 9, 12 months after WBRT, and then every 3 months until date of death from any cause, assessed up to 24 months
  Evaluate neurocognitive function by a standardized neurocognitive battery Trail Making Test Part A & B. TMT-A and B tested the executive function documented with time needed for complete test with no upper limit of range. The longer the time needed, the worse executive function patients preserved.
Neurocognitive function by a standardized neurocognitive battery Controlled Oral Word Association Test | at 1, 2, 4, 6, 9, 12 months after WBRT, and then every 3 months until date of death from any cause, assessed up to 24 months
  Evaluate neurocognitive function by a standardized neurocognitive battery Controlled Oral Word Association Test. Patients are given one phoneme at a time and instructed to say aloud as many words beginning with that phoneme as they could within 1 minute, for a total of three phonemes in 3 minutes. The more the words patients able to say in limit time, the better outcome presented.
Patient reported outcome (Quality of Life questionnaire) | at 1, 2, 4, 6, 9, 12 months after WBRT, and then every 3 months until date of death from any cause, assessed up to 24 months
  EORTC Quality of Life-Core 30 questionnaire module (at question 1 to 27, range from 1 to 4; at question 29 and 30, range from 1 to 7) Quality of Life questionnaire-Brain.
Patient reported outcome (Cognitive Functioning questionnaire) | at 1, 2, 4, 6, 9, 12 months after WBRT, and then every 3 months until date of death from any cause, assessed up to 24 months
  Function Assessment Cancer Therapy for patients with Cognitive function issue
Acute toxicity (Common Toxicity Criteria for Adverse Events version 4) | From date of WBRT until 90 days after radiotherapy starts
  Common Toxicity Criteria for Adverse Events version 4
Late toxicity (Common Toxicity Criteria for Adverse Events version 4) | From 90 days after WBRT starts until the date of death from any cause, up to 60 months
  Common Toxicity Criteria for Adverse Events version 4
Intracranial progression (Number of participant with intracranial progression on MRI of brain) | From date of enrolment until the date of first documented intracranial progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participant with intracranial progression on MRI of brain
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
  Number of patients died

OTHER OUTCOMES:
Genomic risk of neurocognitive decline after WBRT | At 4 months after radiotherapy
  Number of participants with Genomic risk of neurocognitive impairment after WBRT

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No